CLINICAL TRIAL: NCT01170923
Title: Standard Chemotherapy Strategy Versus Changing Chemotherapy Strategy as to FDG-PET Response After 1st Cycle of Standard Chemotherapy for Advanced Non-small Cell Lung Cancer
Brief Title: FDG-PET Scan Response Guided Chemotherapy Strategy for Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sang-We Kim, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMC 08-351
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non small cell lung cancer; FDG PET
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FDG-PET guided (Experimental): Chemotherapy regimen will be changed depending on metabolic response.
  Interventions: Device: FDR-PET
- CT guided (Active Comparator): Chemotherapy regimen will be changed depending on CT findings (RECIST).
  Interventions: Device: CT

INTERVENTIONS:
Device: FDR-PET — FDR-PET performed after 1 cycle of chemotherapy
  Arms: FDG-PET guided
Device: CT — CT performed after 3 cycles of chemotherapy
  Arms: CT guided

SUMMARY:
The usual response to chemotherapy is decided through the image change by computed tomography (CT), which is taken at least 6-9 weeks.

In order to predict the response to chemotherapy earlier, patients received FDG-PET scan at the first cycle of chemotherapy. Chemotherapy was guided by the metabolic response by FDG-PET scan.

DETAILED DESCRIPTION:
Prospective, Open-label, Randomized phase II, single institution trial that compared chemotherapy guided by traditional evaluation based on RECIST versus chemotherapy guided by FDG-PET (metabolic) response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell carcinoma.
2. Stage IIIB (wet) or IV advanced NSCLC.
3. No evidence of prior malignancies for 3 years except treated basal cell or squamous cell carcinoma of skin and carcinoma in situ of uterine cervix.
4. Measurable disease by RECIST criteria.
5. Adequate organ function as follows.

   * Seum AST/ALT < 2.5 x Upper normal limit (UNL) (if hepatic metastasis < 5 x UNL)
   * Total bilirubin < 1.5 x UNL
   * Serum creatinine < 1.5 mg/dL
   * Absolute neutrophil count > 1500/uL
   * Platelet > 100,000/uL
   * Hemoglobin > 9.0 g/dL
6. ECOG Performance status 0-1 7 Age > 18

8. If previously treated with major surgery, it should be over at least 4 weeks. And if previously treated with radiotherapy, it should be over at least 2 weeks.

9. Written consent

Exclusion Criteria:

1. Previous chemotherapy.
2. Symptomatic brain metastasis.
3. Concurrent severe medical illness.
4. Pregnancy and lactation.
5. If there are findings which may increase risk with chemotherapy or inhibit to analyze the result of clinical trial.

   * Uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
change in response rate | within 4 cycles
  The usual response rate of GenexolPM/Cisplatin chemotherapy is 30-40%. This trial will assess whether the changing chemotherapy strategy using FDG-PET can increase response rate by 15%.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-We Kim, MD, Principal Investigator — Asan Medical Center